CLINICAL TRIAL: NCT02084160
Title: The Prediction Value of the BreathID 13C-Methacetin Breath Test for Hepatic Decompensation; a Retrospective Analysis
Brief Title: Prediction Value of the BreathID 13C-Methacetin Breath Test for Hepatic Decompensation
Status: Completed | Type: Observational
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HIS-FU-EX-1213
Record Dates: First submitted 2014-03-09; First posted 2014-03-11 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CLD from HIS-EX-408/PLT-BID-1108: Chronic liver disease subjects from previous Exalenz trial "HIS-EX-408" and PLT-BID1108

SUMMARY:
The objectives of this study are:

* To evaluate the ability of the Methacetin Breath Test (MBT) to detect hepatic decompensation events
* To evaluate the relationship between liver Biopsy and clinical outcome and show that the MBT has a better predictive ability of clinical outcome than liver biopsy.
* To evaluate the ability of the MBT to predict each of the individual liver related complications.

DETAILED DESCRIPTION:
Exalenz has previously gathered information in a previous study on patients with chronic liver disease including the methacetin breath test. Several years later, the company wishes to investigate this group of subjects and see retrospectively if the breath test was a predictor of complications related to their liver disease.

ELIGIBILITY:
Inclusion Criteria:

All subjects that aere enrolled in the previous Exalenz trial HIS-EX-408 or PLT-BID-1108

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic liver disease subjects from previous Exalenz trial "HIS-EX-408"
Sampling Method: Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taufick Chori, MD, Principal Investigator — Hadassah Medical Organization
Locations (4):
- United States (3):
  - Henry Ford Health System, Detroit, Michigan
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Commonwealth University, Richmond, Virginia
- Hadassah Medical Origanzation, Jerusalem, Israel

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CLD From HIS-EX-408/PLT-BID-1108
Started | 579
Completed (579 patient records were reviewed for follow up events, only a small portion had events to report) | 579
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were in previous trials NCT: NCT00736840 and NCT01157845
Arm/Group | CLD From HIS-EX-408/PLT-BID-1108
Number analyzed (Participants) | 579
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.55 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237
  Male | 342
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 418
  Israel | 161

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Decompensation Event
Description: Hepatic decompensation is defined as the occurrence of at least one of the following events in the time frame between the last 13C Methacetin Breath Test (MBT) to the time of data collection:
  1. Death (liver related)
  2. Transplantation (cadaveric and living donors)
  3. Ascites
  4. HE (Hepatic Encephalopathy)
  5. Newly diagnosed varices or variceal bleeding
  6. SBP (spontaneous bacterial peritonitis)
  7. HRS (Hepatorenal syndrome)
  8. HCC (hepatocellular carcinoma)
  9. Increase in CTP (Child Turcotte Pugh) Score by 3 points
  10. Increase in MELD score by 5 points
Time Frame: 5 years
Population: Patients with advanced chronic liver disease
Measure: Number; unit: number of events
Arm/Group | CLD From HIS-EX-408/PLT-BID-1108
Number analyzed (Participants) | 579
number of events | 324

ADVERSE EVENTS:
Time Frame: Not relevant, observational, retrospective
Description: Not relevant, observational, retrospective
Arm/Group | CLD From HIS-EX-408/PLT-BID-1108
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT02084160/Prot_SAP_000.pdf